CLINICAL TRIAL: NCT07152522
Title: Association Between Neck Disability Index Categories and Multidirectional Range of Motion in Patient With Cervical Radiculopathy: Insights From a Cross-Sectional Study
Brief Title: Association Between Neck Disability Index Categories and Multidirectional Range of Motion in Patient With Cervical Radiculopathy
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aida Amir Nassif Naguib, Lecturer of physical therapy, Basic Science department, Cairo University
Other Study IDs: FPTBSUREC/0505/2325
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Cervical Radiculopathy
Keywords: cervical range of motion; neck disability index; cervical radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- cervical radiculopathy with not affected NDI
  Interventions: Other: cross sectional observational
- cervical radiculopathy with mild NDI
  Interventions: Other: cross sectional observational
- cervical radiculopathy with moderate NDI
  Interventions: Other: cross sectional observational
- cervical radiculopathy with severe NDI
  Interventions: Other: cross sectional observational

INTERVENTIONS:
Other: cross sectional observational — the therapist measured ROM in six directions: flexion, extension, right and left side bending, and right and left rotation to investigate the association between NDI and ROM of cervical spine

SUMMARY:
This study aims to investigate the association between NDI categories (None, Mild, Moderate, Severe) and ROM in six directions: flexion, extension, right and left side bending, and right and left rotation. Additionally, it seeks to identify which movements are most affected by neck disability and explore their predictive value for overall ROM changes.

DETAILED DESCRIPTION:
Neck pain is a prevalent musculoskeletal condition that affects a significant portion of the population, with substantial implications for daily functioning and quality of life. The Neck Disability Index (NDI) is a widely used tool to assess the severity of neck pain and its impact on functional activities. Understanding how neck disability correlates with physical impairments, such as reduced range of motion (ROM), is crucial for effective diagnosis and management of this condition.

Despite the established relationship between neck pain and functional limitations, there is limited research quantifying the specific impact of varying levels of neck disability on multidirectional ROM. Furthermore, key directions of movement most affected by neck pain remain underexplored, limiting the ability of clinicians to target interventions effectively.

Scope and Limitations This cross-sectional study focuses on ROM measurements and their relationship with NDI categories. While providing valuable insights, it does not assess changes over time or include other factors such as muscle strength or pain intensity. Addressing these aspects in future research can provide a more comprehensive understanding of neck pain and its implications.

This cross-sectional study included 80 patients diagnosed with neck pain. Participants were categorized into four groups based on their Neck Disability Index (NDI) scores: None, Mild, Moderate, and Severe. Inclusion criteria required participants to have chronic neck pain, while individuals with systemic diseases or comorbid conditions affecting mobility were exclude.

Neck range of motion (ROM) was measured in six directions: flexion, extension, right and left side bending, and right and left rotation. ROM was assessed using a standardized goniometer, and all measurements were performed by the same trained examiner to ensure consistency. NDI scores were obtained through a validated self-reported questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Both male & female
2. Aged 25-60
3. BMI 18.5: 25
4. With cervical radiculopathy that persist for more than 3 months

Exclusion Criteria:

1. Prior surgery to the cervicothoracic spine
2. Bilateral symptoms
3. Signs of upper motor neuron impairments
4. Cervical spine injection in the previous 4 weeks
5. Current use of steroidal anti-inflammatory drugs

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will be conducted in the out-patient clinic Faculty of physical therapy, Cairo University. The expected duration to recruit patients and collect data is 6 months .
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
the association between NDI categories (None, Mild, Moderate, Severe) and ROM in six directions: flexion, extension, right and left side bending, and right and left rotation. | 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Giza, Cairo University, Egypt